CLINICAL TRIAL: NCT03613298
Title: Evaluation of the Location and the Treatment by High-intensity Focused Ultrasounds (HIFU) of Posterior Deep Infiltrating Endometriosis (DIE) Lesions With Intestinal Involvement
Brief Title: Treatment by HIFU With Focal One® of Posterior Deep Infiltrating Endometriosis Lesions With Intestinal Involvement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EDAP TMS S.A. (Industry)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/F/13.12
Record Dates: First submitted 2018-07-20; First posted 2018-08-03 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Endometriosis
Keywords: HIFU; High Intensity Focused Ultrasound; DIE; rectal endometriosis; safety profile; Deep invasive endometriosis; Endometriosis, rectum
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU (Focal One®) Treatment (Experimental): Subjects harboring an isolated recto-sigmoid deep invasive endometriosis (DIE) lesion with a persistence of symptoms despite hormonal treatment will be installed on the Focal One® device to:
  * Evaluate its ability to locate and assess the volume of the endometriosic lesion
  * Treat the targeted lesion by HIFU energy application. Real-time guided ultrasonography will be used to determine the location of the endometriosic nodule.
  Patients will fill-out questionnaires on gynecological and intestinal symptoms and on quality of life before treatment and 1 and 6 months after HIFU. Imaging follow-up scans will be organized at 1 and 6 months and by a pelvic MRI scan at 3/6 months.
  Interventions: Device: HIFU (Focal One®)

INTERVENTIONS:
Device: HIFU (Focal One®) — Endometriosic lesion localization and HIFU treatment will be conducted with the Focal One® device. The treatment area will be defined using sonography, pelvic MRI and a transrectal sonography data. Once the pre-defined lesion will be located with Focal One device, succession of HIFU exposure will then be used to treat maximum lesion volume, excluding a security margin of 3 mm with the digestive mucosae.
  Other Names: High-Intensity Focused Ultrasounds

SUMMARY:
Deep invasive endometriosis (DIE) includes lesions of the rectosigmoid. Theses lesions are associated with painful symptoms that can alter quality of life. High Intensity Focused Ultrasound (HIFU) is a non-invasive ablative procedure using a high-intensity ultrasound probe to induce tissue devitalization using acoustic cavitation and thermal ablation. Focal One® is a transrectal HIFU device, which is validated to treat prostatic cancer.

The primary objective of this clinical trial is to evaluate the ability of the Focal One® HIFU device to detect and target posterior DIE lesions with intestinal involvement. The secondary objectives are to perform a HIFU lesion, to evaluate morphological modifications of the nodule in post-therapeutic imaging scans, to assess evolution of gynecological symptoms, intestinal symptoms, and patients' quality of life after treatment by HIFU and to collect safety data.

DETAILED DESCRIPTION:
20 Subjects with deep invasive endometriosis (DIE) will receive the HIFU treatment with Focal One® device.

Subjects harboring an isolated recto-sigmoid DIE lesion with a persistence of symptoms despite hormonal treatment will be installed on the Focal One® device to:

* Evaluate its ability to locate and assess the volume of the endometriosic lesion
* Treat the targeted lesion by HIFU energy application. Real-time guided ultrasonography will be used to determine the location of the endometriosic nodule. Succession of HIFU exposure will be then used to treat maximum lesion volume, excluding a security margin of 3 mm with the digestive mucosae to prevent risk of fistulae.

Patients will fill-out questionnaires on gynecological and intestinal symptoms and on quality of life before treatment and at 1 and 6 months after HIFU procedure. Imaging follow-up scans will be organized at 1 and 6 months and by a pelvic MRI scan at 3/6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 25 years
* Isolated recto-sigmoid DIE lesion, with no other endometriosis location on imaging examination (intestinal, urinary or ovarian), the persistence of symptoms despite hormonal treatment and therefore consideration for surgical management.
* Localization of endometriosic lesion described by US, confirmed by MRI
* Negative urinary pregnancy test and No intention to get pregnant during the following 6 months
* Affiliated to the French Social Security System

Exclusion Criteria:

* Hormonal treatment of endometriosis by Luteinizing Hormone Releasing Hormone agonist (LHRH analogs) of less than 3 months
* Breastfeeding female
* Uro-genital infection in progress (the infection has to be treated before HIFU treatment)
* Anatomical abnormality of the rectum
* Anterior surgery at the level of the anus or rectum
* Presence of an implant (stent, catheter, contraceptive implant) located less than 1 cm from the treatment area.
* History of intestinal inflammatory pathology
* Allergy to latex
* Female with a medical contraindication on MRI
* Female with a medical contraindication to Sonovue® injection
* Female not able to understand the objectives of the study
* Legal person protected by law

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — deep invasive endometriosis (DIE)
Enrollment: 20 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Targeting of the endometriosic lesion | Day 1
  The main criterion of evaluation will lie on the targeting of the Endometriosic lesion with the Focal One® probe.
  Measure of the volume of the Endometriosic lesion to treat: targeted volume (estimation from the measures of the length, the height and the width of the nodule).

SECONDARY OUTCOMES:
Anatomical position of the Focal One probe | Day 1
  The objective is to evaluate the position of the probe within the rectum before HIFU treatment.
Effect of HIFU treatment on endometriosic lesion | Day 1
  Ratio calculation between targeted volume and treated volume and Evaluation of HIFU on symptomatology
Safety of the procedure: assessment of complications during the procedure attributable to the technique | Day 1
  Complications during HIFU treatment attributable to the HIFU energy deposit or the Focal One are described here.
Assessment of Adverse Events during the 6 months follow-up attributable to the technique | 6 months
  Complications post HIFU treatment.
Medical Outcome assessment (Study Short Form-36) | 6 months
  self-administrated questionnaire: French version of the 36-item Short Form Survey (SF-36)
endometriosis health profile assessment | 6 months
  self-administrated questionnaire: endometriosis health profile (EHP-5)
Urinary symptom profile assessment | 6 months
  self-administrated questionnaire: urinary symptom profile (USP)
Sexual function assessment | 6 months
  self-administrated questionnaire: Female Sexual Function Index (FSFI)
Constipation assessment | 6 months
  self-administrated questionnaire: Knowles-Eccersley-Scott-Symptom Questionnaire (KESS score)
Anal continence assessment | 6 months
  self-administrated questionnaire: Wexner score of anal continence

CONTACTS AND LOCATIONS:
Overall Officials: Gil DUBERNARD, MD PhD, Principal Investigator — Hôpital de la Croix Rousse Service de Gynécologie-Obstétrique, Hospices Civils de Lyon, 103, Grande rue de la Croix Rousse 69 004 Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No